CLINICAL TRIAL: NCT06368362
Title: The Effectiveness and Mediators of Cognitive Bias Modification for Interpretation in the Reduction of Negative Emotional Response to Pain in Individuals With Chronic Musculoskeletal Pain
Brief Title: Cognitive Bias Modification for Interpretation Individuals With Chronic Musculoskeletal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBM-I001
Record Dates: First submitted 2024-04-04; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Chronic Pain; Musculoskeletal Pain Disorder
Keywords: Cognitive bias modification; Interpretation bias
MeSH Terms: conditions — Chronic Pain; Collagen Diseases

STUDY DESIGN:
Intervention Model Description: Two groups of participants (chronic musculoskeletal pain, healthy) were recruited, and within each group participants were randomised to one of two experimental conditions with a 1:1 allocation ratio with a parallel design. Participants with chronic musculoskeletal pain were randomised to benign CBM-I or no CBM-I, and healthy participants were randomised to benign CBM-I or pain-related CBM-I.
Who Masked: Participant
Masking Description: Participants are not informed of the conditioned they are randomised to in this psychological intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Benign CBM-I - Chronic pain (Experimental): Chronic pain participants randomised to receive benign CBM-I, which uses the Ambiguous Situations Task to train participants to neutral meanings of ambiguous scenarios.
  Interventions: Behavioral: Benign cognitive bias modification for interpretation
- No CBM-I - Chronic pain (No Intervention): Chronic pain participants randomised to the 'no CBM-I' condition complete the Ambiguous Situations Task without any form of bias modification.
- Benign CBM-I - Healthy (Experimental): Healthy participants randomised to receive benign CBM-I, which uses the Ambiguous Situations Task to train participants to neutral meanings of ambiguous scenarios.
  Interventions: Behavioral: Benign cognitive bias modification for interpretation
- Pain-related CBM-I - Healthy (Other): Healthy participants randomised to receive pain-related CBM-I, which uses the Ambiguous Situations Task to train participants to painful meanings of ambiguous scenarios.
  Interventions: Behavioral: Pain-related cognitive bias modification for interpretation

INTERVENTIONS:
Behavioral: Benign cognitive bias modification for interpretation — Benign cognitive Bias Modification for Interpretation (CBM-I) trains participants to interpret ambiguous information as neutral or benign rather than pain-related.
  Arms: Benign CBM-I - Chronic pain; Benign CBM-I - Healthy
Behavioral: Pain-related cognitive bias modification for interpretation — Pain-related cognitive Bias Modification for Interpretation (CBM-I) trains participants to interpret ambiguous information as pain-related.
  Arms: Pain-related CBM-I - Healthy

SUMMARY:
Cognitive Bias Modification for Interpretation (CBM-I) trains participants to interpret ambiguous information as neutral or benign, rather than interpret it as being related to pain. The goal of this randomised controlled trial was to explore the feasibility and potential clinical benefits of CBM-I in people with chronic pain and also healthy, pain-free individuals.

DETAILED DESCRIPTION:
This study investigated whether Cognitive Bias Modification for Interpretation (CBM-I) could reduce negative emotional response to pain and to pain-related images, and whether reductions in interpretation bias (IB) and fear of pain mediated this effect. Participants with chronic musculoskeletal pain (N = 41) were randomised to benign CBM-I or no CBM-I, and healthy participants (N = 41) were randomised to benign CBM-I or pain-related CBM-I. After CBM-I, the study assessed pain-related IB and fear of pain, as well as negative emotional response to exercise-induced pain and images of musculoskeletal pain.

ELIGIBILITY:
Chronic pain group Inclusion criteria

* Experience musculoskeletal pain (pain in muscles, bones, joints, tendons, or ligaments) that has lasted for at least the last 3 months before enrolment in the study
* Have visited a healthcare professional for their pain
* Aged 18-70 years
* Normal or corrected to normal vision
* Fluency in the English language Exclusion criteria
* Any known reading difficulty

Healthy group Inclusion criteria

* Aged 18-70 years
* Normal or corrected to normal vision
* Fluency in the English language Exclusion criteria
* Experience frequent or continuous pain for the past three months before enrolment in the study
* Currently experiencing pain
* Any known reading difficulty

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Emotional response to exercise induced pain | Immediately post-intervention
  Sensory and emotional pain words from the McGill Pain Questionnaire (MPQ) were presented, grouped as they are on the MPQ. Participants chose one word from each group most representing the pain experienced performing a dynamic arm exercise (rotating their arms in small circles forwards for 10 seconds then backwards for 10 seconds, repeating the process as many times as possible).
  Participants rated each word from 0 (not at all representative) to 10 (extremely representative) or indicated if none represented their exercise pain. Emotional response to exercise pain was calculated from intensity and representativeness scores. For intensity, words were assigned a numeric score according to MPQ instructions and summed for emotional and sensory words. For representativeness, mean rating of representativeness was calculated for sensory and emotional pain words. The sensory score was subtracted from the emotional score to compute emotional response to pain relative to the sensory experience.
Emotional response to pain-related images | Immediately post-intervention
  Participants were presented twenty pain-related images, and asked to rate the extent to which they felt negative emotions while viewing the image. After a fixation cross presented for 500 ms, a pain-related picture was presented for 6000 ms. This was followed by another cross presented for 500 ms then numbers from 0 (not at all negative) to 10 (very negative) was displayed. Participants were instructed to look at the picture on the screen then to rate their negative emotion from 0 (not at all negative) to 10 (very negative). The mean rating of emotional response to pain-related images was calculated for each participant.

SECONDARY OUTCOMES:
Fear of Pain | Immediately post-intervention
  Fear of Pain Questionnaire - III. A 30-item scale (0 - Not at all, to 5 - Extreme), including three subscales: major pain (e.g., a car accident), minor pain (e.g. biting your tongue), and medical pain (e.g. an injection), with 10 items in each subscale. Higher scores indicate higher levels of pain-related fear.
Anxiety | Baseline
  Anxiety subscale of the Hospital Anxiety and Depression Scale (HADS). A seven-item subscale of the 14-item HADS (ranging from 0 - 3, or 3 - 0), with higher scores indicating higher levels of anxiety.
Depression | Baseline
  Depression subscale of the Hospital Anxiety and Depression Scale (HADS). A seven-item subscale of the 14-item HADS (ranging from 0 - 3, or 3 - 0), with higher scores indicating higher levels of depression.
Emotional response to average clinical pain | Immediately post-intervention
  Sensory and emotional pain words from the McGill Pain Questionnaire (MPQ) were presented, grouped as they are on the MPQ. Participants chose one word from each group that was most representative of their average experience of clinical musculoskeletal pain. Participants rated each word on a scale from 0 (not at all representative) to 10 (extremely representative), or indicated if none of the words were representative of their pain. Indices of emotional response to musculoskeletal pain were calculated from intensity and representativeness scores. For intensity, words were assigned a numeric score according to the MPQ scoring instructions and these were summed for emotional and sensory words separately. For representativeness, the mean rating of representativeness was calculated for sensory and affective/evaluative (emotional) pain words separately. The sensory score was subtracted from the emotional score to determine the emotional response to pain relative to the sensory experience.
Pain severity | Baseline
  Pain severity subscale of the Brief Pain Inventory - Short Form, assessing pain at its worst and least in the last 24 hours, on average, and right now on a scale of 0 (no pain) to 10 (pain as bad as you can imagine).
Pain interference | Baseline
  Pain interference subscale of the Brief Pain Inventory - Short Form. A seven-item subscale which assesses the extent to which pain has interfered with general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life over the past 24 hours on a scale of 0 (does not interfere) to 10 (completely interferes).
Pain-related interpretation bias index | Immediately post-intervention
  Assessed via Ambiguous Scenarios Task. The training phase presents ambiguous scenarios with a fragment of the last word shown, which participants completed. In the pain-related modification condition, the final word gave the scenario a pain-related meaning. In the benign modification condition, the final word gave the scenario a neutral meaning. The test phase assesses whether participants interpret new ambiguous scenarios as pain-related or benign, with participants rating the similarity of four endings (two pain-related and two neutral) to the original scenario from 1 (very different in meaning) to 4 (very similar in meaning). The mean score for benign target endings was subtracted from the mean score for negative endings to give an index of interpretation bias (a positive index indicates pain-related interpretation bias). To assess visual imagery, participants rated how easily they could imagine themselves as the protagonist in the scenarios from 1 (not at all) to 5 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Schoth, PhD, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant dataset that underlies the results reported in this article may be requested from the authors.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Twelve months following publication of the results.
Access Criteria: Email the study authors.